CLINICAL TRIAL: NCT03555643
Title: Evaluation of the Hyperintense Acute Reperfusion Marker for the Detection of a Cerebral Ischemia in the Anterior and Posterior Circulation in Patients With Transient Ischemic/Neurological Attack
Brief Title: Evaluation of the HARM for the Detection of a Cerebral Ischemia in TIA/TNA Patients
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Alex Förster, MD, Universitätsmedizin Mannheim
Other Study IDs: 2016-591N-MA
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: TIA; Stroke; Ischemia; Diagnoses Disease
Keywords: TIA; Stroke; Ischemia; MRI; FLAIR; hyperintense acute reperfusion marker
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transient ischemic attack (TIA): Patients with transient ischemic attack
- transient neurological attack (TNA): Patients with transient neurological attack

SUMMARY:
The research project investigates the incidence of the hyperintense acute reperfusion marker (HARM) in patients with transient ischemic attack (TIA) or transient neurological attack (TNA). Initially, HARM was described after acute ischemic stroke and is caused by a blood-brain barrier disorder after recanalization of an acute vessel occlusion and consecutive reperfusion. These result in a contrast agent extravasation into the subarachnoid space, which can be easily detected on fluid attenuated inversion recovery (FLAIR) images.

TIA is defined as a transient focal neurological deficit with a probably cerebrovascular cause. In contrast, TNA is defined as a transient non-focal neurological deficit with multiple causes, including cerebrovascular. The clinical diagnosis of TIA is often flawed and the delineation of TIA and TNA can be difficult. MRI is the most important diagnostic method for the detection or exclusion of cerebral ischemia in patients with TIA/TNA in daily clinical practice. However, on diffusion-weighted imaging (DWI) approximately two-thirds of TIA cases and only one-fifth of TNA cases demonstrate acute cerebral ischemia. Supplementary perfusion-weighted imaging (PWI) scans can only slightly increase this percentage. The well-known HARM could prove to be complementary to DWI and PWI and close or at least reduce the existing gap. In the case of TNA in particular, this could be of clinical relevance in order to avoid mistreatment or even dismissal without further clarification after supposedly inconspicuous imaging.

Therefore, the aim of this study is to record the incidence of HARM in a statistically significant number of cases of patients with TIA and TNA and to investigate relationships with symptom duration and anatomical localization. In addition, the dynamics of contrast enhancement in the subarachnoid space in TIA and TNA cases with HARM will be analyzed in detail.

ELIGIBILITY:
Inclusion Criteria:

* transient focal neurological symptoms (aphasia, facial paresis, hemiparesis, hemihypaesthesia, double vision, hemianopia, hemiataxia, etc.)
* transient non-focal neurological symptoms (confusion, dizziness, memory deficits, gait insecurity, bilateral weakness, etc.)
* MRI examination possible within 24 hours of symptoms
* able to give informed consent

Exclusion Criteria:

* persistent symptoms
* symptoms lasting more than > 24 h
* clinical suspicion of other cause of symptoms (seizures, intoxication, hypoglycemia, psychogenic)
* contraindications for MRI (pacemaker, metallic splinter, cochlear implants, etc.)
* unable to give consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (≥ 50 years) with transient focal or non-focal neurological symptoms who are eligible for an MRI examination within 24 hours after onset of symptoms and able to give informed consent.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
hyperintense acute reperfusion marker (HARM) | within 24 hours after onset of symptoms
  Detection of the hyperintense acute reperfusion marker (HARM) on postcontrast FLAIR images.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Förster, MD, Principal Investigator — Universitätsmedizin Mannheim, Dept. of Neuroradiology
Locations (1):
- Universitätsmedizin Mannheim, Mannheim, Germany